CLINICAL TRIAL: NCT07212283
Title: Wise Intervention for Reducing Aggressive Behaviors and Promoting Prosocial Behaviors Toward LGB-TNB Individuals
Acronym: LGB-TNB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Deusto (Other)
Responsible Party: Principal Investigator, Nerea Cortazar Enciondo, PhD, University of Deusto
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ETK-90/24-25
Record Dates: First submitted 2025-09-30; First posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-09

CONDITIONS: Aggression; Adolescence
Keywords: Adolescence; LGBTQ; Aggression; Prosocial Behavior; Wise Intervention
MeSH Terms: conditions — Aggression; Altruism

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial with two groups will be used. Randomization will be done by clusters, using the classroom as the unit. First, the schools will be selected according to their characteristics. Then, half of the participants will be assigned to the experimental intervention (condition 1) and the other half to the control intervention (condition 2) in parallel for the duration of the study.
Who Masked: Participant, Outcomes Assessor
Masking Description: Allocation will be concealed to the participants and teachers. Assessment will be done online through self-reports.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Values alignment wise intervention (Active Comparator)
  Interventions: Behavioral: Values alignment wise intervention
- Wise Intervention LGB-TNB (Experimental)
  Interventions: Behavioral: Wise Intervention LGB-TNB

INTERVENTIONS:
Behavioral: Wise Intervention LGB-TNB — The intervention will be designed to reduce aggressive behaviors based on sexual orientation and gender identity and to promote prosocial behaviors toward these individuals. This intervention will include three components: (1) reading scientific studies about people's ability to change. In addition, they will read other studies about how thoughts and emotions influence behavior through brain pathways, and that these pathways can be modified under certain circumstances; (2) reading testimonials that support the idea that people can change. These testimonials include accounts of people who were victims or perpetrators based on sexual orientation and gender identity, including important components of empathy and prosocial behaviors toward the victims. To give credibility to the intervention, they will be informed that these stories were written by other young people who previously participated; and (3) self-persuasion exercises that involve an active commitment to change.
  Arms: Wise Intervention LGB-TNB
Behavioral: Values alignment wise intervention — This intervention will be based on the same strategies as the experimental intervention, but it will not address aspects related to prosocial behaviors or aggression toward LGB-TNB individuals; instead, it will be applied to improve adolescents' eating habits.
  Arms: Values alignment wise intervention

SUMMARY:
This study evaluates the effectiveness of a wise Intervention to reduce aggressive behaviors and promote prosocial behaviors toward LGB-TNB individuals among Spanish adolescents. Half of the participants will receive the experimental intervention, while the other half will receive a control intervention.

DETAILED DESCRIPTION:
Discrimination based on sexual orientation and gender identity is a social problem of great relevance. Sexual orientation is understood as the mechanism that directs affective-sexual attraction and interest, manifesting with varying intensity. Regarding gender identity, it has historically been interpreted under a binary paradigm based on external sexual organs, rendering trans and non-binary identities invisible. However, it is currently understood as the internal feeling about one's own gender, so that trans and/or non-binary people represent those whose gender identity differs from the one assigned at birth.

Despite the growing visibility, public awareness, and recognition of the rights of lesbian, gay, bisexual, trans, and non-binary people (LGB-TNB), discrimination based on sexual orientation and gender identity continues to be a social problem of great relevance with serious consequences for those who suffer it. This reality underlines the need to implement effective interventions aimed at addressing these aggressive behaviors and the mechanisms that sustain them, not only among those who perpetrate acts of violence, but also among people who witness these aggressive behaviors.

In addition, intervening during adolescence is especially relevant, as this stage represents a critical moment in the moral, social, and emotional development of individuals. Moreover, during adolescence, discriminatory behaviors and peer aggression increase, and previous studies show that LGB-TNB people face a higher risk of violence in educational settings. Nevertheless, although adolescence becomes a critical period for the development of risk behaviors, it also involves important transitions and learning opportunities. Furthermore, adolescence is a turning point during which well-designed interventions have a high potential to redirect a person's developmental trajectory in a lasting way. Therefore, it can be an especially favorable moment for implementing interventions.

In this way, numerous interventions have been carried out in educational settings to prevent aggressive behaviors among peers. Although most of these initiatives have mainly focused on more general problems, such as bullying and cyberbullying, in recent years preventive interventions specifically aimed at reducing aggressive behaviors based on sexual orientation and gender identity in both face-to-face and digital contexts have increased. However, most current interventions focus on educating people about issues related to LGB-TNB topics, reaching mixed and contradictory results regarding their effectiveness, and also highlighting that there is little empirical evidence about the robustness of the effects of LGB-TNB interventions and their underlying mechanisms. Therefore, these interventions present areas for improvement that constitute important challenges for scientific psychology.

Recently, interest has grown in social psychology regarding a new approach to interventions, which have been called wise interventions. Many of these interventions have impactful results because they are usually very brief in time and produce lasting changes in people's behavior. Moreover, this type of intervention is of great interest in adolescence, as they allow themselves to be designed in such a way that they are perceived as respectful of students' autonomy and status, so that they feel they are making their own decisions.

Therefore, the aim of this project is to adapt to the LGB-TNB context a wise intervention to reduce online and offline aggression among adolescents, especially based on sexual orientation and gender identity, and to increase the intention to support and prosocial behaviors when participants witness these aggressions, especially those directed at LGB-TNB people.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent by the adolescents and their families.
* To be fluent in Spanish and/or Euskera.

Exclusion Criteria:

* Lack of permission by families and the adolescent.
* Lack of understanding of the instructions.

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1000 (Estimated)
Dates: Start 2025-09-18 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in aggression scores toward LGB-TNB individuals, assessed using an adaptation of the Spanish version (Orue et al., 2018) of the Homophobic Bullying Scale (Prati, 2012). | Assessments were conducted at baseline and at 3, 6, and 9 months.
  It consists of seven items that ask frequency with wich participants have engaged in specific aggressive behavior toward LGB-TNB individuals. Five response categories are provided using a Likert-type response scale, ranging from 1 (never) to 5 (daily).
Change from baseline in online aggression scores toward LGB-TNB individuals, assessed using the Technology-Facilitated Gender- and Sexuality-Based violence (TFGSV; Martínez-Bacaicoa et al., 2023). | Assessments were conducted at baseline and at 3, 6, and 9 months.
  It consists of eight items that ask frequency with wich participants have engaged in online aggressive behavior toward LGB-TNB individuals. Five response categories are provided using a Likert-type response scale, ranging from 1 (never) to 5 (daily).
Change from baseline in prosocial behavior scores toward LGB-TNB individuals through an ad hoc measure. | Assessments were conducted at baseline and at 3, 6, and 9 months.
  It consists of one item in which participants were asked to select all the behaviors they engaged in after witnessing an aggression.
Change from baseline in bystander intention scores when witnessing aggressive behavior toward LGB-TNB individuals. | Assessments were conducted at baseline, immediately after the intervention, and at 3, 6, and 9 months.
  This measure evaluate bystander intentions in response to LGB-TNB aggressions, through different scenarios. After reading the scenarios, participants answered five items that evaluated possible courses of action to take in response to the aggression.

SECONDARY OUTCOMES:
Change from baseline in moral disengagement scores, assessed using the mechanisms of moral disengagement described by Bandura (2016) and based on studies with similar characteristics (Martínez-Bacaicoa et al., 2024). | Assessments were conducted at baseline and at 3, 6, and 9 months.
  It consists of eight items representing the eight mechanisms that allow participants to morally disengage. Five response categories are provided using a Likert-type response scale, ranging from 1 (strongly disagree) to 5 (strongly agree).
Change from baseline in justice sensitivity scores, assessed using the Justice Sensitivity Inventory (Schmitt et al., 2010). | Assessments were conducted at baseline and at 3, 6, and 9 months.
  It consists of 10 items that assess sensitivity to unjust situations. Five response categories are provided using a Likert-type response scale, ranging from 1 (strongly disagree) to 5 (strongly agree).
Change from baseline in behaviors supporting LGB-TNB individuals, assessed using the LGBT-Affirming Behavior questionnaire (Poteat, 2015). | Assessments were conducted at baseline and at 3, 6, and 9 months.
  It consists of five items that assess supportive behaviors toward LGB-TNB individuals. Five response categories are provided using a Likert-type response scale, ranging from 1 (0 times) to 5 (7 or more times).
Change from baseline in microaggression scores toward LGB-TNB individuals, assessed using the Sexual Orientation Microaggression Scale (SOMS-P; Botor & Tuliao, 2025) and the Gender Identity Microaggression Scale (GIMS-P; Botor & Tuliao, 2025). | Assessments were conducted at baseline and at 3, 6, and 9 months.
  A total of 25 items are used to assess microaggressions toward LGB-TNB individuals. Specifically, 20 items assess microaggressions toward LGB individuals and 5 items assess microaggressions toward TNB individuals. Five response categories are provided using a Likert-type response scale, ranging from 1 (never) to 5 (almost every week).
Change from baseline in offline perpetration scores, assessed using the Spanish adaptation (Ortega-Ruiz et al., 2016) of the European Bullying Intervention Project Questionnaire (Brighi et al., 2012). | Assessments were conducted at baseline and at 3, 6, and 9 months.
  It consists of six items that ask about the frequency with which participants have engaged in aggressive behaviors in offline contexts. Five response categories are provided using a Likert-type response scale, ranging from 1 (never) to 5 (almost every week).
Change from baseline in online perpetration scores, assessed using an adaptation of the Cyberbullying Questionnaire items (Calvete et al., 2010; Gámez-Guadix et al., 2014). | Assessments were conducted at baseline and at 3, 6, and 9 months.
  It consists of five items that ask about the frequency with which participants have engaged in aggressive behaviors in online contexts. Five response categories are provided using a Likert-type response scale, ranging from 1 (never) to 5 (almost every week).
Change from baseline in healthy and unhealthy food intake scores, assessed using an adaptation of the KIDMED 2.0 questionnaire, validated in a sample of Spanish children and adolescents (López-Gajardo et al., 2022). | Assessments were conducted at baseline and at 3, 6, and 9 months.
  It consists of 16 items that ask about the frequency of healthy and unhealthy food intake. Five response categories are provided using a Likert-type response scale, ranging from 1 (never) to 5 (daily).
Change from baseline in alignment of healthy eating habits scores, as assessed by the questionnaire developed by Bryan et al. (2019). | Assessments were conducted at baseline, immediately after the intervention, and at 3, 6, and 9 months.
  It consists of seven items that assess the alignment between participants' healthy eating habits and their personal values. Five response categories are provided using a Likert-type response scale, ranging from 1 (strongly disagree) to 5 (strongly agree).

CONTACTS AND LOCATIONS:
Locations (1):
- Nerea, Bilbao, BIZKAIA, Spain

IPD SHARING:
Plan to Share IPD: Yes
Raw data will be available at OSF when the results of the study are published.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The study protocol and informed consent protocol will be published at clinicaltrials.org. Data will be available at OSF when the results are published.
Access Criteria: Public

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-09-25): https://cdn.clinicaltrials.gov/large-docs/83/NCT07212283/Prot_SAP_000.pdf
  • Informed Consent Form (2025-09-25): https://cdn.clinicaltrials.gov/large-docs/83/NCT07212283/ICF_001.pdf